CLINICAL TRIAL: NCT03189433
Title: Phase 2, Multiple-Site, Open-Label, Randomized, 2-Group, Parallel Study to Assess the Efficacy and Safety of Ryanodex(R) (EGL-4101)as Adjuvant Treatment in Subjects With Psychostimulant Drug-Induced Toxicity (PDIT)
Brief Title: Efficacy and Safety Study of Ryanodex as Adjuvant Treatment in Subjects With Psychostimulant Drug-Induced Toxicity (PDIT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited enrollment
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGL-4104-C-1702
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-11

CONDITIONS: Drug Toxicity Psychotropic Agents Psychostimulants
MeSH Terms: interventions — Dantrolene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ryanodex + Standard of Care (Active Comparator): Ryanodex (dantrolene sodium) 50 mg/mL suspension to be administered as a rapid IV push of 2.5 mg/kg, added to Standard of Care (SOC). SOC is defined as efficient body cooling by physical methods and supportive measures [ice packs, evaporative cooling(application of room temperature water via mist with use of a fan], benzodiazepines to ameliorate shivering, IV fluids, respiratory support, and other treatments deemed necessary to treat complications or comorbidities]. Administer a single dose of Ryanodex. If a subject does not show an adequate clinical response within 10 - 30 minutes post-dose, a second IV bolus dose of 2.5 mg/kg may be administered.
  Interventions: Drug: Ryanodex (dantrolene sodium) for injectable suspension
- Standard of Care only (SOC) (No Intervention): Standard of Care is defined as efficient body cooling by physical methods and supportive methods and supportive measures[ice packs, evaporative cooling (application of room temperature water via mist with use of a fan], benzodiazepines to ameliorate shivering, IV fluids, respiratory support, and other treatments deemed necessary to treat complications or comorbidities].

INTERVENTIONS:
Drug: Ryanodex (dantrolene sodium) for injectable suspension — Ryanodex (dantrolene sodium) for injectable suspension, 250 mg/vial to be reconstituted in 5 mL of sterile water for injection to yield a 50 mg/mL suspension that will be administered as a rapid IV push of 2.5 mg/mL.
  Arms: Ryanodex + Standard of Care

SUMMARY:
Ryanodex is being investigated as a potential adjuvant treatment for people suffering from psychostimulant drug-induced toxicity (PDIT), a life-threatening medical condition that results mainly from the abuse of certain illicit drugs, most notably methamphetamine, and related forms (MDMC or "Molly"; MDMA or "Ecstasy"). Ryanodex is approved for the treatment of malignant hyperthermia in conjunction with appropriate supportive measures and for prevention of malignant hyperthermia in patients at high risk and in this study, will be investigated for the treatment of PDIT. The hypothesis of this study is that administration of Ryanodex as adjuvant treatment to Standard of Care (SOC) will improve the clinical outcome compared with SOC alone, in subjects with psychostimulant drug induced toxicity. Current SOC is defined as body cooling and supportive measures.

DETAILED DESCRIPTION:
This study will be conducted at pre-hospital emergency care (PHEC) facilities. The PHECs are medical units that are fully equipped and staffed to provide adequate emergency medical care to patients with PDIT. The study is designed to evaluate the safety and efficacy of Ryanodex in an on0site pre-hospital emergency setting where subjects are anticipated to be treated over a short period of time and then transferred to another medical facility or released. After screening and diagnosis of PDIT, SOC treatment will be initiated. Subjects eligible for the study will be randomized to either receive SOC + Ryanodex or to receive SOC only. Study subjects are expected to remain at the study site for a maximum of 6 hours post-baseline.

ELIGIBILITY:
Inclusion Criteria: Male and non-pregnant subjects diagnosed with psychostimulant drug induced toxicity as evidenced by all of the following: core body temperature of greater than or equal to 39.5 degrees C; organ dysfunction, as evidenced by a Logistic Organ Dysfunction System score of greater than or equal to 6 (In the event of any delay in obtaining the results for baseline LODS score determination, subject may be enrolled. After enrollment, if the pending baseline LODS score turns out to be less than 6, the subject will be withdrawn from the study and replaced); known or suspected us of a psychostimulant drug in the judgment of the Investigator; negative blood pregnancy test for females (in the event of any delay in obtaining pregnancy test result, subject may be enrolled and randomized if all of the other eligibility criteria are met).

Exclusion Criteria: Diagnosed with or is suspected to have an acute, clinically severe infection, which may, in the opinion of the Investigator, may increase the subject's risk for participating in the study an/or may impair the ability of performing and/or interpreting study assessments; severe hyperthermia secondary to a condition other than a psychostimulant drug-induced toxicity; likelihood of head trauma in the past 3 months, or other systemic disease that might increase the subject's risk for participating in the study and/or may impair the ability of performing and/or interpreting study assessments; positive pregnancy test or evidence of active lactation; known history of allergy or hypersensitivity to dantrolene; known history of seizure disorders or epilepsy; current or prior use (within the past 2 weeks) of calcium channel blockers.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CrowdRx Medical Office- Moonrise Festival, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ryanodex + Standard of Care | Standard of Care Only (SOC)
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: No patients were entered in the SOC group
Groups:
- Total: Total of all reporting groups
Arm/Group | Ryanodex + Standard of Care | Standard of Care Only (SOC) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieved a Logistic Organ Dysfuction System (LODS) Total Score Less Than or Equal to 5
Description: Logistic Organ Dysfunction System (LODS) score (measure/scoring of 1-3 specific parameters in 6 organ systems; neurologic, cardiologic, renal, pulmonary, hematologic, and hepatic). One to 5 LODS points are assigned to the levels of severity and the resulting LODS scores range can range from 0 to 22 points. A lower score represents a better outcome; a score of 0 points is a better outcome than a score o 22 points.
Time Frame: At or prior to 60 minutes post-randomization
Population: Due to lack of enrollment, data was insufficient for a meaningful analysis. Data were not collected.
Arm/Group | Ryanodex + Standard of Care | Standard of Care Only (SOC)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Subjects Who Achieved a LODS Total Score Less Than or Equal to 5 at Other Planned Time Points.
Description: Proportion of subjects who achieved a LODS total score less than or equal to 5 at other planned time points. One to 5 LODS points are assigned to the levels of severity and the resulting LODS scores range can range from 0 to 22 points. A lower score represents a better outcome.
Time Frame: Up to 6 hours post-dose.
Population: Data were not collected and thus could not be analyzed.
Arm/Group | Ryanodex + Standard of Care | Standard of Care Only (SOC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: NA: No adverse event data were collected; time frame is 0 hours, 0 days, 0 months.
Description: Adverse events were not monitored/assessed.
Arm/Group | Ryanodex + Standard of Care | Standard of Care Only (SOC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Pi is not permitted to discuss or publish trial results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03189433/SAP_000.pdf
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03189433/Prot_001.pdf